CLINICAL TRIAL: NCT01393106
Title: A Phase 2 Study to Assess the Efficacy and Safety of GS-1101 (CAL-101) in Patients With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: Safety and Efficacy of Idelalisib in Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101-11
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2015-11

CONDITIONS: Hodgkin Lymphoma
Keywords: HL; idelalisib; CAL-101; GS-1101; PI3K
MeSH Terms: conditions — Hodgkin Disease | interventions — idelalisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Idelalisib (Experimental): Participants will receive up to 300 mg of idelalisib twice daily.
  Interventions: Drug: Idelalisib

INTERVENTIONS:
Drug: Idelalisib — Idelalisib tablets administered orally
  Other Names: Zydelig®; GS-1101; CAL-101

SUMMARY:
This study will evaluate the efficacy and safety of idelalisib in participants with relapsed of refractory Hodgkin Lymphoma (HL). The primary objective will be to assess the overall response rate.

Eligible participants will initiate oral therapy with idelalisib at a starting dose of 150 mg twice daily. Treatment with idelalisib will continue until tumor progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years
* Karnofsky performance score of ≥ 60 (Eastern Cooperative Oncology Group (ECOG) performance score of 0, 1, or 2)
* Histologically confirmed diagnosis of classic HL (ie, nodular sclerosis, mixed cellularity, lymphocyte depleted, and or lymphocyte rich types)
* Nodal HL that shows fluorodeoxyglucose (FDG) avidity (defined as focal or diffuse FDG uptake above background in a location incompatible with normal anatomy or physiology), and is measurable (defined as the presence of ≥ 1 nodal lesion that measures ≥ 2 cm in a single dimension as assessed by CT, PET/CT, or magnetic resonance imaging (MRI))
* Relapsed or refractory HL after prior myeloablative therapy with autologous stem cell transplantation (ASCT) or after ≥ 2 prior chemotherapy-containing regimens and no curative option with conventional therapy
* Discontinuation of all radiotherapy or chemotherapy for the treatment of HL greater than or equal to 3 weeks before initiation of study treatment and discontinuation of all radioimmunotherapy for HL (Visit 2)
* All acute toxic effects (excluding alopecia, neurotoxicity, or anemia) of any prior antitumor therapy resolved to Grade ≤ 2 before initiation of study treatment (Visit 2)
* For men and women of childbearing potential willingness to abstain from sexual intercourse or employ an effective method of contraception during the study drug administration and follow-up periods
* Willingness and ability to provide written informed consent and to comply with protocol requirements

Exclusion Criteria:

* Known active central nervous system or leptomeningeal lymphoma
* History of a non-lymphoma malignancy except for the following: adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, localized prostate cancer, other adequately treated Stage 1 or 2 cancer currently in complete remission, or any other cancer that has been in complete remission for ≥ 5 years
* Evidence of ongoing systemic bacterial, fungal, or viral infection (excluding viral upper respiratory tract infections) at the time of initiation of study treatment (Visit 2)
* Pregnancy or breastfeeding
* Ongoing alcohol or drug addiction
* Known history of drug-induced liver injury, chronic active hepatitis C virus (HCV), chronic active hepatitis B virus (HBV), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, ongoing extrahepatic obstruction caused by stones, cirrhosis of the liver or portal hypertension
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing immunosuppressive therapy, including systemic corticosteroids.
* Prior therapy with idelalisib
* Exposure to another investigational drug within 3 weeks prior to start of study treatment
* Concurrent participation in another therapeutic treatment trial
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, ECG finding, or laboratory abnormality that, in the investigator's opinion, could affect the safety of the patient; alter the absorption, distribution, metabolism or excretion of the study drug; or impair the assessment of study results
* Prior therapy with any drug that inhibits Akt, Bruton tyrosine kinase (BTK), Janus kinase (JAK), mammalian target of rapamycin (mTOR), phosphatidylinositol 3 kinase (PI3K) (including idelalisib), or spleen tyrosine kinase (SYK)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndah Dreiling, MD, Study Director — Gilead Sciences
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Gopal AK, Fanale MA, Moskowitz CH, Shustov AR, Mitra S, Ye W, Younes A, Moskowitz AJ. Phase II study of idelalisib, a selective inhibitor of PI3Kdelta, for relapsed/refractory classical Hodgkin lymphoma. Ann Oncol. 2017 May 1;28(5):1057-1063. doi: 10.1093/annonc/mdx028. PMID 28327905

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 15 September 2011. The last study visit occurred on 28 August 2014.
Pre-assignment Details: 32 participants were screened.
Groups:
- Idelalisib: Idelalisib up to 300 mg (75, 100, or 150 mg tablets) administered orally twice daily until tumor progression or development of unacceptable toxicity.
Period: Overall Study
Arm/Group | Idelalisib
Started | 25
Completed | 20 (Completed: Disease Progression/Death)
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Analysis Set: participants who received at least one dose of study drug.
Arm/Group | Idelalisib
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 1
  Black or African American | 2
  White | 19
  Other | 3
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
Time Since Diagnosis (years) [Mean (Standard Deviation); unit: years] | 3.9 (4.26)
Classical Hodgkin Lymphoma Pathologic Subtype [Number; unit: participants]
  Nodular Sclerosis | 23
  Lymphocyte Rich | 2
Disease Stage at Screening [Number; unit: participants] — Disease stage was based on the Ann Arbor Lymphoma Staging System:
  Stage I: Single lymph node group or lymph node region; Stage II: Two or more node regions on same side of diaphragm; Stage III: Lymph node regions on both sides of the diaphragm; Stage IV: Multiple extranodal sites or lymph nodes and extranodal sites
  participants
    Stage I | 1
    Stage II | 8
    Stage III | 6
    Stage IV | 10
Karnofsky Performance Status [Mean (Standard Deviation); unit: units on a scale] — Classifies patients according to their functional impairment. Scores range from 0-100; the lower the score, the worse the survival for most serious illnesses.
  units on a scale | 83 (7.1)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) was assessed based on the International Working Group Revised Response Criteria for Malignant Lymphoma (Cheson, 2007), and was defined as the proportion of participants achieving a complete response (CR) or partial response (PR) as assessed by the investigator.
  * CR was defined as the complete resolution of all disease-related radiological abnormalities and the disappearance of all signs and symptoms related to the disease.
  * PR was defined as a ≥ 50% reduction in the sum of the products of the longest perpendicular diameters of all index lesions, with no new lesions.
Time Frame: Up to Week 110
Population: Intent-to-treat (ITT) Analysis Set: participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 25
percentage of participants | 20.0 [6.8 to 40.7]

2. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the interval from the first documentation of PR or CR to the earlier of the first documentation of disease progression or death from any cause.
Time Frame: Up to Week 110
Population: Responding Analysis Set: participants who achieved a best response of CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib
Number analyzed (Participants) | 5
months | 8.4 [1.8 to NA] — Not reached

3. Secondary Outcome: Percent Change From Baseline in the Sum of the Product of the Greatest Perpendicular Diameters (SPD) of Target Lymph Nodes as Documented Radiographically
Time Frame: Baseline, Week 8, Week 48, and up to Week 110
Population: ITT Analysis Set
Measure: Median (Full Range); unit: percent change in SPD
Arm/Group | Idelalisib
Number analyzed (Participants) | 25
percent change in SPD
  Percent Change at Week 8 (n = 24) | -14.1 [-73.1 to 112.5]
  Percent Change at Week 48 (n = 5) | -45.9 [-92.6 to 7.8]
  Best Percent Change from Baseline (n = 24) | -24.1 [-92.6 to 112.5]

4. Secondary Outcome: Change From Baseline in Fluorodeoxyglucose (FDG) Uptake in Lymph Nodes as Assessed by Positron-emission Tomography (PET)
Time Frame: Up to Week 110
Population: An analysis of changes in FDG uptake by the tumor was not conducted due to unavailability of lymph node biopsy samples.
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Response
Description: Time to response (TTR) was defined as the interval from the start of idelalisib treatment to the first documentation of CR or PR.
Time Frame: Up to Week 110
Population: Responding Analysis Set
Measure: Median (Full Range); unit: months
Arm/Group | Idelalisib
Number analyzed (Participants) | 5
months | 2.0 [1.9 to 16.8]

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from start of idelalisib treatment to death from any cause.
Time Frame: Up to Week 110
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib
Number analyzed (Participants) | 25
months | 19.8 [12.3 to NA] — Not reached

7. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) was defined as the interval from the start of idelalisib treatment to the earlier of the first documentation of disease progression or death from any cause.
Time Frame: Up to Week 110
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Idelalisib
Number analyzed (Participants) | 25
months | 2.3 [1.8 to 3.7]

8. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure (TTF) was defined as the interval from the start of idelalisib treatment to the earlier of the first documentation of disease progression, the permanent cessation of idelalisib therapy due to an adverse event, or death from any cause.
Time Frame: Up to Week 110
Population: No data are presented because time to treatment failure data were not collected.
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

9. Secondary Outcome: Changes in Health-related Quality of Life as Reported Using the Functional Assessment of Cancer Therapy: Lymphoma (FACT-Lym) Questionnaire
Description: Change in health-related quality of life was reported by participants using the FACT-Lym questionnaire assessment tool. Results are presented as the mean (SD) best change from baseline in FACT-Lym total score, which was defined as the highest change score (improvement) after baseline.
  The FACT-Lym total score is on a scale from 0-168, with higher scores associated with a better quality of life.
Time Frame: Baseline and up to Week 110
Population: FACT-Lym Evaluable Analysis Set: participants who had sufficient baseline and on-study measurements to provide interpretable results for this endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Idelalisib
Number analyzed (Participants) | 20
units on a scale | 5.1 (7.24)

10. Secondary Outcome: Changes in Performance Status as Documented Using the Karnofsky Performance Criteria for Participants ≥ 16 Years of Age and the Lansky Performance Criteria for Participants < 16 Years of Age
Description: Changes in performance status were assessed using the Karnofsky performance criteria for participants ≥ 16 years of age and the Lansky performance criteria for participants < 16 years of age. Since there were no participants < 16 years of age, only the Karnofsky performance criteria were used. The change in Karnofsky performance status was reported as the best (highest change score) and worst (lowest change score) change from baseline using the Karnofsky performance criteria. The Karnofsky score classifies patients according to their functional impairment. Scores are on a scale from 0-100, the lower the score, the worse the survival for most serious illnesses.
Time Frame: Baseline and up to Week 110
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Idelalisib
Number analyzed (Participants) | 7
units on a scale
  Best Change | 6 (5.3)
  Worst Change | -1 (6.9)

11. Secondary Outcome: Changes in the Plasma Concentrations of Disease-associated Chemokines and Cytokines
Time Frame: Up to Week 110
Population: This analysis was not conducted due to discrepancies with the transfer of samples.
Arm/Group | Idelalisib
Number analyzed (Participants) | 0

12. Secondary Outcome: Overall Safety Profile of Idelalisib
Description: The overall safety of idelalisib was assessed as the percentage of participants experiencing adverse events (AEs; Serious AEs, Grade ≥ 3 AEs, AEs related to idelalisib, and AEs leading to discontinuation of idelalisib), clinically significant abnormal electrocardiograms (ECG), and laboratory abnormalities. "Clinically significant" abnormalities in ECG were as determined by the investigator.
Time Frame: Up to Week 110
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Idelalisib
Number analyzed (Participants) | 25
percentage of participants
  Any AE | 96.0
  Serious AE | 36.0
  Grade ≥ 3 AE | 48.0
  AE related to idelalisib | 76.0
  AE leading to permanent drug discontinuation | 8.0
  Clinically significant abnormal ECG at Week 16 | 0
  Grade 3 or 4 hemoglobin | 4.0
  Grade 3 or 4 neutrophils | 8.0
  Grade 3 or 4 platelets | 4.0
  Grade 3 or 4 alanine aminotransferase | 20.0
  Grade 3 or 4 aspartate aminotransferase | 16.0

13. Secondary Outcome: Compliance With Study Drug Dosing as Assessed by Accounting for Used and Unused Drug
Time Frame: Up to Week 110
Population: ITT Analysis Set
Measure: Mean (Standard Deviation); unit: number of doses
Arm/Group | Idelalisib
Number analyzed (Participants) | 25
number of doses
  Number of doses dispensed | 463 (462.3)
  Number of doses taken | 329 (321.1)

14. Secondary Outcome: Idelalisib Trough and Peak Plasma Concentration at Week 4
Description: Plasma samples were collected predose (trough) and 1.5 hours postdose (peak). The minimum and maximum value among participants sampled at each time point are presented. Results of less than the lower limit of quantitation (ie, 5 ng/mL) were treated as zero prior to the achievement of the first quantifiable concentration and as missing otherwise.
Time Frame: Predose and 1.5 hours postdose at Week 4
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Number; unit: ng/mL
Arm/Group | Idelalisib
Number analyzed (Participants) | 25
ng/mL
  Trough - minimum (n = 20) | 142
  Trough - maximum (n = 20) | 2120.0
  Peak - minimum (n = 22) | 90.2
  Peak - maximum (n = 22) | 8570.0

ADVERSE EVENTS:
Time Frame: Up to Week 110
Description: ITT Analysis Set
Arm/Group | Idelalisib
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=25)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Herpes zoster (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Platelet count decreased (Investigations) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hospitalisation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib (N=25)
Anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Tachycardia (Cardiac disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 6
Chills (General disorders) | 5
Fatigue (General disorders) | 8
Pain (General disorders) | 2
Pyrexia (General disorders) | 6
Upper respiratory tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 5
Aspartate aminotransferase increased (Investigations) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Memory impairment (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
There were no limitations affecting the analysis or results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years